CLINICAL TRIAL: NCT01217684
Title: Test-retest Reliability of a Standard Protocol on the Biodex Dynamometer
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML 6404
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Test-retest Reliability; Validity; Biodex Medical Systems III Dynamometer; Experimental Measure of Knee Extension Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of the present study is to evaluate test-retest reliability of a standard protocol on the Biodex dynamometer in older adults.

In addition, the test-retest reliability and validity of an experimental measure of knee extension strength will be assessed in older adults.

ELIGIBILITY:
Inclusion Criteria:

* +65 years old
* able to perform a maximal strength test on a dynamometer

Exclusion Criteria:

* pathologies that prohibit a maximal strength test on a dynamometer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older adults
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Leuven, Belgium